CLINICAL TRIAL: NCT03369093
Title: Efficacy of Two Doses of Parenteral Amoxicillin Plus Single Dose Gentamicin Compared to Four Doses of Parenteral Ampicillin Plus Single Dose Gentamicin in Managing Children Hospitalized With WHO Classified Severe Pneumonia: a RCT
Brief Title: RCT of Efficacy of Amoxicillin Over Ampicillin on Severe Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR-17061
Record Dates: First submitted 2017-09-25; First posted 2017-12-11 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Treatment Failure; Lethargy; Altered Mental Status; Convulsion, Non-Epileptic; Hypoxia; Feeding; Difficult, Newborn
Keywords: RCT; severe pneumonia; amoxicillin; under five
MeSH Terms: conditions — Lethargy; Seizures; Hypoxia; Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Investigators have completed the enrollment of 308 participants by the study endline. All the Serious adverse events have been reported appropriately to the Ethical Review Committee and the Data Safety and Monitoring Board (DSMB)
Who Masked: Participant
Masking Description: This was an unblinded intervention trial. Blinding could not be justified by the ethical review committee as the schedule of administration of the drugs was different and drug dispensing-related side effects were investigators' other concern.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ampicillin arm (Active Comparator): Ampicillin arm: Patients will receive four doses of parenteral Ampicillin and single dose of Gentamicin daily for 3-5 days
  Interventions: Drug: Amoxicillin
- Amoxicillin arm (Experimental): Amoxicillin arm: Patients will receive two doses of Amoxicillin and single dose of Gentamicin daily for 3-5 days
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Twice daily doses of injectable amoxicillin
  Other Names: no other intervention

SUMMARY:
Burden: Pneumonia remains the leading infectious cause of death accounting for 920,000 children under five around the world. This means a loss of over 2,500 child lives every day, or over 100 every hour. Since 2000, the number of child deaths caused by pneumonia has decreased by 47 percent. The tremendous progress made is due in part to the rapid roll-out of vaccines, better nutrition, and improved care-seeking and treatment for symptoms. However, pneumonia hasn't declined as quickly as other diseases such as malaria (58%), HIV/AIDS (61%), and measles (85%).

Knowledge gap: The Lancet Series on Childhood Pneumonia and Diarrhea has reported that case management is one of the three most effective interventions to reduce pneumonia deaths in children. It is also noted that the cost-effectiveness of these interventions in the national health system needs urgent assessment. It was suggested to find out means to reduce hospital stay without compromising the quality of care.

Relevance: The main purpose of the study is to compare the efficacy of two doses of parenteral Amoxicillin plus single-dose Gentamicin compared to four doses of parenteral Ampicillin plus single-dose Gentamicin. After 72 hours of treatment injectable Amoxicillin or injection Ampicillin will be switched to or replaced by oral Amoxicillin and will be discharged with an advice to attend to Ambulatory Care Unit (ACU) to receive a once-daily dose of injection Gentamicin for a total of 5 days. It is anticipated that this modified therapy will reduce the hospitalization stay of children with severe pneumonia and would therefore be relevant in countries with the resource-poor settings. By reducing the hospitalization period, this therapy has the potentials to reduce hospital-acquired infection.

Hypothesis (if any): Rate of treatment failure with two doses of injectable Amoxicillin plus single-dose Gentamicin will be no more than that of four doses of injectable Ampicillin plus single-dose Gentamicin in the management of children between 2 months to 59 months hospitalized for WHO classified severe pneumonia.

DETAILED DESCRIPTION:
Severe pneumonia is a serious infection in children which requires timely intervention. Management of severe pneumonia is done by appropriate antibiotics and supportive care. WHO recommendation is to use injection ampicillin four times a day for 3-5 days and injection gentamicin once a day for 3-5 days in children with severe pneumonia. In the study, the investigators want to compare the response of injection ampicillin with another similar and equally effective antibiotic (amoxicillin). The reason for choosing amoxicillin is that the dose is two times a day and it is cost-effective and reduces chances of nosocomial infection. The response of the drugs will be compared by the time difference of clinical improvement of the patients or time difference of disappearance of the sign and symptoms on admission. The investigators are interested to compare the recovery time from the illness as well as treatment failure in both groups. In that way, the investigators will be able to develop a better treatment for pneumonia in children in low-cost settings.

The study will be an open-label, randomized, controlled intervention in children between two months to 59 months admitted to Dhaka Hospital of icddr,b. Investigators will use sealed envelopes to randomly assign the children to either treatment arm. In the first arm children will receive 2 daily doses of parenteral Amoxicillin and a single daily dose of parenteral Gentamicin; and in 2nd arm, children will receive 4 daily doses of parenteral Ampicillin and a single daily dose of parenteral Gentamicin. After 72 hours of treatment, injection Amoxicillin and injection Ampicillin will be replaced with oral Amoxicillin but injection gentamicin will be continued for a total of 5 days in one daily dose. During this time participants will be suggested to discharge from the hospital and attain to the Ambulatory care unit for getting a once-daily dose of injection of Gentamicin. Both the treatment arm will continue for 5 days.

During the study period, participants in both study arms will also receive standardized hospital management for other co-morbidities-such as diarrhea, malnutrition, and any other complications. Hypoxia will be managed by B-CPAP through a nasal cannula.

Any participants will be declared "Treatment failure" who show the persistence of danger signs after 48 hours or develop new danger signs within 24 hours of initiation of antibiotic treatment. If a participant needs mechanical ventilation, dies at any time during a hospital stay, or left the hospital against medical advice will be also declared as a treatment failure.

Participants from either study group who develops the features of "treatment failure" should be rescued with the second-line antibiotic regimen, which is injection ceftriaxone and injection levofloxacin.

Monitoring of the children with severe pneumonia The following parameters should be routinely monitored in every child with severe pneumonia. Special attention should be given to participants receiving I/V fluid therapy and those with SAM. Such as: Heart rate, respiratory rate, temperature, respiratory pattern including chest recession, lower chest wall indrawing, use of accessory muscles, the establishment of oral feeding, liver size, oxygen saturation level, chest auscultation: (rales, rhonchi, bilateral basal crepitation, pleural rub), fluid and calorie intake.

Participants on oxygen therapy should have at least 3-4 hourly observations of all the above parameters and participants without getting oxygen should be observed at least 2 hourly by the study nurses. All the patients should be evaluated by the physicians at least 12 hourly.

Signs of Improvement:

In absence of complications, within 2 days of initiation of treatment, there should be signs of improvement i ) breathing rate within normal limit; ii) absence of the lower chest wall in-drawing; iii) less to no fever; iv) improved ability to eat and drink, and v) better oxygen saturation without assistance.

Discharge criteria

* Respiratory distress has resolved
* Oxygen saturation > 90%
* Feeding well
* Able to take oral medication or have completed a course of parenteral antibiotics
* The parents understand the signs of pneumonia, risk factors, and when to return

The study objective is to compare the efficacy of two doses of injectable Amoxicillin plus single-dose injectable Gentamicin compared to four doses of injectable Ampicillin plus single-dose injectable Gentamicin in the management of participants hospitalized with WHO pneumonia.

Secondary objectives are to compare time to resolution of danger signs of pneumonia, length of hospital stay, mortality rate, rate of complication requiring mechanical ventilation, and rate of multiorgan or renal or cardiac failure between the two treatment groups.

Children more than 2 months to less than 59 months will be enrolled in the study, if participants have a history of cough or difficulty in breathing and WHO classified severe pneumonia plus at least two of the following:

i) Central cyanosis or oxygen saturation <90% on pulse oxymetry ii) Severe respiratory distress (e.g. grunting, very severe chest indrawing) iii) Signs of pneumonia with a general danger sign: inability to breastfeed or drink; lethargy or reduced level of consciousness; convulsion iv) In addition, some or all of the other signs of pneumonia may be present, such as:

* Signs of pneumonia [age specific fast breathing( Annex 1)]
* Chest indrawing: lower chest wall indrawing
* Chest auscultation signs: (any one)

  1. Decreased breath sounds
  2. Bronchial breath sounds
  3. Crackles
  4. Abnormal vocal resonance (decreased over a pleural effusion or empyema, increased over lobar consolidation)
  5. Pleural rub

Participants with a life-threatening condition that required immediately assisted ventilation or referring to an outside hospital (such as septic shock, cardiac arrest, apnea, respiratory failure, etc.) will be excluded from the study. Children with uncorrected cyanotic CHD, hypercapnia (PCO2 > 60mm of Hg), status asthmaticus and upper-airway obstruction, preterm baby (but not ex-preterm), and those for who inform consent can't be secured from their parents/ care-givers. Caregivers presented with any drug container of antibiotics or prescription showing getting antibiotics will be excluded.

Sample size calculation:

[For two-sample comparison of proportion (non-inferiority)]

Null hypothesis: p2-p1≤ δ (inferior), where: pi (entered in command) is the overall proportion of participants expect to experience the outcome of the treatments are non-inferior, and delta is the smallest change in proportions between groups (p2 - p1) which would still be clinically important.

Assumptions:

power = 0.8; alpha = 0.025 (one-sided); pi = 0.50; delta = 0.16 Estimated required sample size (per group) = 154,

Total sample is 308

This study will be conducted at the Dhaka Hospital of icddr,b, Dhaka, Bangladesh. This hospital is located in Dhaka city, the capital of Bangladesh. It provides care and treatment to around 110,000 diarrheal patients with or without associated complications and with or without other health problems each year. The vast majority of the patients come from poor socio-economic backgrounds from urban and peri-urban Dhaka, the capital city of Bangladesh.

Patients attending this hospital are first assessed by an experienced triage nurse, which includes assessment of the type of diarrhea and degree of dehydration, and presence of other health problems including ALRI/ pneumonia, severe malnutrition, impaired mental status (convulsion), and sepsis. The non-diarrhoeal patients have been redirected to other appropriate hospitals in the city. Based on an assessment of diarrhoeal patients, those with uncomplicated illness without signs of dehydration are referred to the Out-Patient Department (OPD) for 4-5 hours of observation, maintenance of hydration using ORS solution, and for provision of health education to the mothers/caregivers. Those with some and severe dehydration but without any associated health problems are admitted to Short Stay Ward (SSW) for correction of dehydration and maintenance of hydration using ORS and/or intravenous fluids, provision of antimicrobial therapy as appropriate, with an average stay of 24 hours. Those with associated complications of diarrhea and/or associated health problems are referred to a physician for assessing the need for admission to either the Longer Stay Ward (LSW) or Acute Respiratory Ward (ARI) or to the Intensive Care Word (ICU) depending on the clinical severity. The usual associated conditions include difficult respiration, cyanosis, apnoea, hypothermia or hyperthermia, marked lethargy or comatose condition, poor peripheral perfusion not attributable to severe dehydration. Participants hospitalized in SSW are assessed by hospital clinicians for possible admission to LSW and further workup and management. After admission to the LSW/ARI/SCU, the attending physician will obtain medical history, performs a thorough clinical examination, makes a problem list including differential diagnoses for each of them, arranges for required laboratory workups, and develops the treatment plan following standard guidelines of the hospital. Investigators will also perform bedside procedures such as sampling blood, performing lumbar punctures, etc. Oxygen saturation is determined by pulse oximeter when necessary, and blood glucose estimated by bedside Gluco Check machine in nearly all patients admitted to the LSW/ARI /SCU.

ELIGIBILITY:
Inclusion Criteria:

1. WHO classified severe pneumonia

Exclusion Criteria:

1. Very sick children require mechanical ventilation
2. Children with any congenital or structural defect

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 308 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment failure | within 48 hours
  Persistence of danger signs of severe pneumonia such as hypoxia, feeding difficulty, abnormal mentation after 48 hours or new appearance of danger sign within 24 hours

SECONDARY OUTCOMES:
Time of resolution or recovery from pneumonia period for pneumonia | 48 hours
  Recovery from features of pneumonia in terms of respiratory distress, abnormal chest auscultation finding
Total length of hospitalization | 3-5 days
  Period of hospitalization
Nosocomial infection | 7 days
  any hospital acquired infection proven by laboratory facility
Post discharge morbidity | 30 days
  Follow up over phone to get information of any mild illness at home after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lubaba Shahrin, MBBS, FCPS, Principal Investigator — Dhaka Hospital
Locations (1):
- Dhaka Hospital, icddr,b, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shahrin L, Chisti MJ, Shahid ASMSB, Rahman ASMMH, Islam MZ, Afroze F, Huq S, Ahmed T. Injectable Amoxicillin Versus Injectable Ampicillin Plus Gentamicin in the Treatment of Severe Pneumonia in Children Aged 2 to 59 Months: Protocol for an Open-Label Randomized Controlled Trial. JMIR Res Protoc. 2020 Nov 2;9(11):e17735. doi: 10.2196/17735. PMID 33136058